CLINICAL TRIAL: NCT07181148
Title: A Prospective, Randomized, Single-blinded (Investigator), Parallel, Multi-center, Active-control, Non-inferiority, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of MSP01-T for Bowel Cleansing Before Colonoscopy
Brief Title: A Study to Evaluate the Safety and Effectiveness of MSP01-T for Bowel Cleansing Before a Colonoscopy
Acronym: MSP01
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mather's Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MTS-P01-2401
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: MSP01-T; Colonoscopy; Colon Cleanse; Oral Bowel Cleanser; Oral Tablet; Randomized Trial; Phase 3 Study

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug Group (Experimental): 2-day split-dose
  Interventions: Drug: MSP01-T
- Control Drug Group (Active Comparator): 2-day split-dose
  Interventions: Drug: MSP01-R

INTERVENTIONS:
Drug: MSP01-R — Total 20 tablets, split-dose administration over 2 days: 14 tablets the day before colonoscopy, 14 tablets on the morning of colonoscopy, oral intake.
  Other Names: Orafang Tab
  Arms: Control Drug Group
Drug: MSP01-T — Total 20 tablets, split-dose administration over 2 days: 10 tablets the day before colonoscopy, 10 tablets on the morning of colonoscopy, oral intake.
  Arms: Test Drug Group

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of MSP01-T, a new bowel cleansing agent, in adults who are scheduled to undergo a colonoscopy.

Participants will be randomly assigned to receive either MSP01-T or a comparator product.

The study will assess how effectively MSP01-T cleans the bowel before the procedure and monitor any potential side effects.

Adults aged 19 years and older who are planning to have a colonoscopy may be eligible to take part.

DETAILED DESCRIPTION:
Colonoscopy is a widely used diagnostic and screening procedure for colorectal diseases. Adequate bowel cleansing is essential for the accuracy and safety of the procedure. MSP01-T is a new bowel cleansing agent developed to improve patient compliance and cleansing quality while minimizing side effects.

This phase 3, randomized, single-blind, multicenter, active-controlled, non-inferiority clinical trial is designed to evaluate the efficacy and safety of MSP01-T compared to an existing standard bowel preparation. Participants will be randomly assigned to receive MSP01-T or a comparator product before undergoing a colonoscopy.

The primary objective of this study is to assess the quality of bowel preparation as evaluated by endoscopists using a standardized scoring system. Secondary objectives include patient-reported tolerability, safety assessments including adverse events, and overall satisfaction.

Adults aged 19 years and older who are scheduled for a colonoscopy may be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 19 years or older at the time of providing written informed consent.
2. Individuals scheduled to undergo a screening colonoscopy.
3. 19 kg/㎡ ≤ BMI < 30 kg/㎡
4. Participants who have voluntarily agreed to participate in the clinical trial and have provided written informed consent.

Exclusion Criteria:

Participants who meet any of the following will NOT be eligible to participate in this clinical trial:

1. Colonoscopy for therapeutic purposes, including:

   * Hemostatic treatment after vascular malformation, ulcer, tumor, or polypectomy
   * Decompression for non-toxic megacolon or sigmoid volvulus
   * Foreign body removal
   * Balloon dilation of strictures
   * Palliative treatment for bleeding due to strictures or tumors
2. Medical history at screening, including:

   * Epilepsy or seizure within 2 years
   * Severe cardiac disease within 24 weeks (e.g., unstable angina, acute myocardial infarction)
   * Clinically significant gastrointestinal or abdominal surgery within 24 weeks (except appendectomy, hemorrhoidectomy)
   * Active infection or fever ≥ 38°C within 1 week (except mild upper respiratory infection or localized skin infection)
   * Hypersensitivity to investigational product components
3. Concomitant diseases at screening, including:

   * Active gastrointestinal bleeding
   * Coagulation disorders
   * Gastrointestinal obstruction, perforation, or gastric emptying disorders
   * Inflammatory bowel disease (e.g., Crohn's disease, toxic megacolon, toxic colitis)
   * Acute abdomen requiring surgery
   * Major cardiovascular disease (e.g., congestive heart failure [NYHA class III-IV], clinically significant arrhythmia, QTcF > 450 msec [male] or > 470 msec [female])
   * Uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg)
   * Insulin therapy requirement
   * Clinically significant electrolyte imbalance
   * Risk of dehydration (e.g., rhabdomyolysis, ascites)
   * Severe renal impairment (eGFR < 30 mL/min/1.73 m²)
   * ALT or AST > 3 × ULN
   * Severe nausea or vomiting interfering with trial participation
   * Active hepatitis B (HBsAg positive) or hepatitis C (HCV Ab positive)
   * HIV positive
   * Neurological or psychiatric disorders (e.g., depression, bipolar disorder, epilepsy, substance abuse) or use of related medications
4. Medication use:

   * Severe constipation (bowel movement < 3/week) or regular use of laxatives/prokinetics within 12 weeks
   * Use of laxatives, enemas, simethicone, 5-HT4 agonists, iron, or opioids within 7 days before Day 1
5. Pregnant or breastfeeding women
6. Women of childbearing potential and men unwilling to use effective contraception during the study
7. Participation in another clinical trial and receipt of investigational drug or device within 4 weeks
8. Any condition judged inappropriate by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with "successful" bowel cleansing based on HCS [by independent central reader] | During colonoscopy
  Percentage of participants assessed as having "successful" bowel preparation by independent central reader based on Harefield Cleansing Scale (HCS). "Successful" = HCS grade A or B.

SECONDARY OUTCOMES:
Proportion of participants with "successful" bowel cleansing based on HCS [by investigator] | During colonoscopy
  Percentage of participants assessed as having "successful" bowel preparation by investigator based on Harefield Cleansing Scale (HCS). "Successful" = HCS grade A or B.
Overall bowel cleansing score based on HCS [by independent central reader] | During colonoscopy
  Proportion of participants, as assessed by an independent central reader, classified as grade A, B, C, or D based on the Harefield Cleansing Scale (HCS), which evaluates the quality of bowel cleansing. Overall bowel cleansing is considered "successful" if graded A or B, and "unsuccessful" if graded C or D.
Overall bowel cleansing score based on HCS [by investigator] | During colonoscopy
  Proportion of participants, as assessed by the investigator, classified as grade A, B, C, or D based on the Harefield Cleansing Scale (HCS), which evaluates the quality of bowel cleansing. Overall bowel cleansing is considered "successful" if graded A or B, and "unsuccessful" if graded C or D.
Segmental bowel cleansing scores (5 colonic segments) based on HCS [by independent central reader] | During colonoscopy
  HCS score for each of 5 colonic segments assessed by independent central reader. Each of the five colonic segments is scored on a 5-point scale (0-4) as follows:
  0 = Irremovable, heavy, hard stools;
  1. = Semi-solid, only partially removable stools;
  2. = Brown liquid, removable semi-solid stools;
  3. = Clear liquid;
  4. = Empty and clean. Scores of 3 or 4 are considered "high quality cleansing."
Segmental bowel cleansing scores (5 colonic segments) based on HCS [by investigator] | During colonoscopy
  Same as above, but assessed by the site investigator. Each of the five colonic segments is scored on a 5-point scale (0-4) as follows:
  0 = Irremovable, heavy, hard stools;
  1. = Semi-solid, only partially removable stools;
  2. = Brown liquid, removable semi-solid stools;
  3. = Clear liquid;
  4. = Empty and clean. Scores of 3 or 4 are considered "high quality cleansing."
Proportion of participants with residual bubbles based on Bubble Score [by independent central reader] | During colonoscopy
  Proportion of participants with a bubble score of ≥1, as assessed on a 4-point scale (0-3) for overall and segmental evaluation (Grade 0: No or minimal scattered bubbbles, Grade 1: Bubbles covering at least half the luminal diameter, Grade 2: Bubbles covering the circumference of the lumen, Grade 3: Bubbles filling the entire lumen).
Proportion of participants with residual bubbles based on Bubble Score [by investigator] | During colonoscopy
  Same as above, but assessed by the site investigator.
Proportion of participants with detected polyps or adenomas [by investigator] | During colonoscopy
  Participants in whom polyps or adenomas were detected during colonoscopy.
Proportion of participants with cecal intubation achieved [by investigator] | During colonoscopy
  Proportion of participants in whom the colonoscope successfully reached the cecum during colonoscopy
Colonoscopy insertion time [by investigator] | During colonoscopy
  Time from rectal insertion of the colonoscope to confirmation of the cecal base.
Colonoscopy withdrawal time [by investigator] | During colonoscopy
  Time from cecum to anus during colonoscopy withdrawal.
Total colonoscopy procedure time [by investigator] | During colonoscopy
  Total time calculated as the sum of colonoscopy insertion time (from rectal insertion to cecal confirmation) and withdrawal time (from cecal confirmation to removal of the colonoscope from the anus)
Study drug administration satisfaction - Difficulty (score) | Immediately after study drug administration
  Participants rate difficulty of taking study drug on a 5-point Likert scale (1 = very easy, 5 = very difficult); higher scores indicate greater difficulty.
Study drug administration satisfaction - Taste (Score) | Immediately after study drug administration
  Participants rate taste of study drug on a 4-point scale (1 = good, 4 = bad)
Proportion of participants by study drug acceptability | Immediately after study drug administration
  Proportion of participants willing to use the same colon cleansing agent for a future colonoscopy: Yes / No.
Proportion of participants by study drug adherence/compliance | Immediately after study drug administration
  Proportion of participants by total study drug intake: 100%, ≥75% to <100%, <75%.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No